CLINICAL TRIAL: NCT01998555
Title: Development and Evaluation of a Web-based Group Cognitive-behavioral Therapy Program for Coronary Artery Heart Disease Patients
Brief Title: Web-based Psychological Intervention to Coronary Artery Heart Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201306066RINC
Record Dates: First submitted 2013-10-18; First posted 2013-12-02 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAD-CBT group therapy (Other): CAD receive web-based CBT group therapy
  Interventions: Other: CBT
- CAD-CBT group therapy waiting list (Other): CAD waiting list will receive web-based CBT group therapy later
  Interventions: Other: CBT

INTERVENTIONS:
Other: CBT

SUMMARY:
The purpose of this study is to evaluate medical cost-effectiveness, reduce the psychological risk factors( including hostility, anxiety, depression, and perceived stress) in coronary artery disease (CAD) patients and enhance the regulation of the autonomic nervous system (including respiration rate, heart rate, distal blood vessel pulse, and finger temperament) through web-based cognitive -behavioral group therapy.

DETAILED DESCRIPTION:
Cognitive-behavioral therapy (CBT) is effective in reducing the level of anger, hostility and depression present in coronary artery disease (CAD) patients.In Taiwan, Weng et al. also confirmed the eight-week group CBT program not only diminished the emotion disturbances including anger, hostility and depression of CAD, but also significantly prolonged the coagulation time, thus reducing the rate of thrombosis formation. Even though the therapeutic effect of the CBT program was valid, this program is still not accessible for some patients in need because they are not aware of it, or they are restricted by time and transportation. Internet-based therapeutic intervention can overcome the obstacles to access this program at any time and in any place. Presently, structured CBT intervention is provided through the Internet and used widely by patients with physical or psychological problems such as smoking, obesity, or headaches, but not by CAD patients. Therefore, the purpose of this research is to evaluate the effects to reduce the psychological risk factors of a web-based group CBT program in CAD patients. Follow-up assessments will be performed after 3 and 6-month durations. The investigators expect that, after an eight-week group intervention, there will be significant decrease of the psychological risk factors. Moreover, the therapeutic effects can be maintained during the three- and six-month follow-up.evaluate In addition, web-based cognitive -behavioral group therapy will significantly reduce indirect medical costs (travel time and money).

ELIGIBILITY:
inclusion:

1. coronary artery disease
2. regular medication

exclusion:

1.Psychiatric diseases

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Significant decrease of the psychological risk factors in web-based group CBT intervention group after an eight-week group intervention | Time point(s) at post-group intervention, 3 months, and 6 months follow up
  Evaluate the effects to reduce the psychological risk factors and enhance the regulation of automatic nerve system：
  Time point：Post-intervention, 3 months, and 6 months follow up
  Subjective (self report inventories), including hostility, anxiety,and perceived stress.
  Objective (Biofeedback devices):including blood vessel pulse, EKG, skin conductance, ect.

SECONDARY OUTCOMES:
Significantly reduce health care costs | intervention
  Evaluate indirect medical cost-effectiveness (travel time and money) during web-based Psychological Interventions

OTHER OUTCOMES:
Psychosocial risk factor and characteristic cardiovascular responses present present in CAD patients on pre-group intervention | Pre- group intervention
  Time point：Pre-group intervention
  Subjective (self report inventories), including hostility, anxiety,and perceived stress.
  Objective (Biofeedback devices):including blood vessel pulse, EKG, skin conductance, ect.

CONTACTS AND LOCATIONS:
Overall Officials: Bee-Horng Lue, Principal Investigator — National Taiwna University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan